CLINICAL TRIAL: NCT00977691
Title: Nonmyeloablative Haploidentical Peripheral Blood Mobilized Hematopoietic Precursor Cell Transplantation for Severe Congenital Anemias Including Sickle Cell Disease and Beta-Thalassemia
Brief Title: Haploidentical PBMC Transplant for Severe Congenital Anemias
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 090225; 09-H-0225
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Results first posted 2019-10-14 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-12

CONDITIONS: Sickle Cell Anemia
Keywords: Sickle Cell Anemia; Peripheral Blood Stem Cell Transplantation; Graft-Versus-Host Disease; Sirolimus (Rapamune ); Alemtuzumab (Campath ); Thalassemia; Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell; Graft vs Host Disease; Thalassemia | interventions — Alemtuzumab; Sirolimus; Cyclophosphamide; Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): PBSC transplant with no post-transplant cyclophosphamide (PT-Cy)
  Interventions: Procedure: PBSC Transplant; Drug: Alemtuzumab; Drug: Sirolimus; Procedure: Low Dose Irradiation
- Cohort 2 (Experimental): PBSC transplant with 50 mg/kg post-transplant cyclophosphamide (PT-Cy)
  Interventions: Procedure: PBSC Transplant; Drug: Alemtuzumab; Drug: Sirolimus; Drug: Cyclophosphamide; Procedure: Low Dose Irradiation
- Cohort 3 (Experimental): PBSC transplant with 100 mg/kg post-transplant cyclophosphamide (PT-Cy)
  Interventions: Procedure: PBSC Transplant; Drug: Alemtuzumab; Drug: Sirolimus; Drug: Cyclophosphamide; Procedure: Low Dose Irradiation

INTERVENTIONS:
Procedure: PBSC Transplant — PBSC transplant
Drug: Alemtuzumab — alemtuzumab
  Other Names: Campath
Drug: Sirolimus — sirolimus
  Other Names: Rapamune
Drug: Cyclophosphamide — cyclophosphamide
  Other Names: Cytoxan
  Arms: Cohort 2; Cohort 3
Procedure: Low Dose Irradiation — low dose irradiation

SUMMARY:
Background:

Bone marrow transplantation (BMT), which involves transplanting a donor's marrow stem cells, is capable of curing some congenital anemias. BMT usually involves high-intensity treatment with chemotherapy and radiation to kill abnormal cells, which affects all systems of the body.

People with anemias often have damage to other organs such as the kidneys, which can be further damaged by the chemotherapy. Only approximately 20 percent of patients have a full-matched donor, making treatment for many people with anemias unavailable. However, 90 percent of patients may have a half-matched donor, but using a half-matched donor increases the toxicity of BMT.

Objectives:

To determine if a research BMT with half-matched donor cells, low-intensity radiation, immunosuppressant drugs, and no chemotherapy will be effective in patients with sickle cell disease and Beta-thalassemia.

To determine the effectiveness of cyclophosphamide, an immunosuppressant drug, in preventing rejection of the donor cells.

Eligibility:

Recipients are individuals at least 18 years of age who have been diagnosed with sickle cell disease and Beta-thalassemia, and who have a family member who is a haploidentical (i.e., half match) tissue match.

Donors are healthy individuals between the ages of 2 and 80 who are found to be suitable donors.

Design:

Donors will undergo apheresis, which involves withdrawing blood from one arm vein, passing it through a machine that removes bone marrow stem cells, and returning the remaining blood through the vein in the other arm. Donors will receive a drug that causes the stem cells to be released into the bloodstream prior to the apheresis procedure.

Recipients will undergo routine physical and laboratory examinations, including bone marrow sampling at the beginning of the study. After transplantation, physical and laboratory examinations will occur on a weekly or twice weekly basis at the outpatient clinic. Recipients will be examined every 6 months starting 100 days posttransplant for 5 years.

Recipients will receive low-dose radiation in two treatments 1 and 2 days before the transplant. They will also be given immunosuppressant therapy with alemtuzumab and sirolimus. Another immunosuppressant drug, cyclophosphamide, will be given in the future as needed to subsets of the recipients to prevent rejection of donor cells.

Recipients will receive the donor stem cells through a previously inserted central line. The process takes up to 8 hours.

Recipients will receive blood transfusions as necessary to prevent anemia and bleeding during the posttransplant period. They may also receive intravenous antibiotics to prevent infection.

DETAILED DESCRIPTION:
Nonmyeloablative allogeneic peripheral blood stem cell (PBSC) transplants are currently being investigated in phase I/II trials assessing engraftment, efficacy, and toxicity at a number of transplant centers. Our ongoing protocol for patients with severe congenital anemias, particularly sickle cell disease (SCD), and an HLA-matched sibling donor has had excellent preliminary results. None of the patients who engrafted had sickle-related events or any evidence of graft versus host disease (GVHD). There was no significant toxicity associated with the conditioning regimen.

Our main limitation has been a lack of HLA-matched sibling donors in the majority of patients. We performed a study in which patients with severe SCD who lacked a suitable donor underwent a search for a matched unrelated donor or umbilical cord donor. The vast majority of patients were not found to have an appropriate alternative donor. We therefore seek to develop a safe nonmyeloablative regimen to be applied to the haploidentical setting so that family members can serve as donors and greatly expand the donor pool.

In this protocol, we propose PBSC transplantation in patients with SCD and thalassemia, considered at high risk for complications from or ineligible for standard bone marrow transplantation, with allogeneic peripheral blood stem cells from a haploidentical donor using a novel immunosuppressive regimen without myeloablation in an attempt to further decrease the transplant-related morbidity/mortality. The low intensity nonmyeloablative conditioning regimen will consist of a relatively low radiation dose for therapeutic radiation, Alemtuzumab (Campath ), Sirolimus (Rapamune ), and Cyclophosphamide (Cytoxan ) as a strategy to provide adequate immunosuppression to allow sufficient engraftment for clinical remission with a lower risk of GVHD development. T-cell replete, donor-derived, granulocyte colony-stimulating factor (G-CSF)-mobilized PBSC will be used to establish hematopoietic and lymphoid reconstitution.

The primary endpoint of this study is the percentage of patients who have sustained donor type hemoglobin without significant GVHD for patients with SCD, or who are transfusion-independent and without significant GVHD for patients with thalassemia. Other endpoints include degree of donor-host chimerism necessary for long term graft survival and disease amelioration, incidence of acute and chronic GVHD, incidence of graft rejection, transplant-related morbidity, as well as disease-free and overall survival.

ELIGIBILITY:
* INCLUSION CRITERIA:

Recipients (must fulfill one disease category in 5.1.1 and all of 5.1.2)

5.1.1 Disease specific

5.1.1.1 Patients with sickle cell disease (HB SS, SC, or SBeta(0)-thal) at high risk for disease-related morbidity or mortality, defined by having severe end-organ damage (A, B, C, or D) or potentially modifiable complication(s) not ameliorated by hydroxyurea (E):

A. Stroke defined as a clinically significant neurologic event that is accompanied by an infarct on cerebral MRI or cerebral arteriopathy requiring chronic transfusion therapy; OR

B. Sickle cell-related renal insufficiency defined by a creatinine level greater than or equal to 1.5 times the upper limit of normal and kidney biopsy consistent with sickle cell nephropathy OR nephrotic syndrome OR creatinine clearance less than 50mL/min OR requiring peritoneal or hemodialysis; OR

C. Pulmonary hypertension defined as tricuspid regurgitant jet velocity (TRV) of greater than or equal to 2.5 m/s at baseline (without vaso-occlusive crisis); OR

D. Sickle hepatopathy defined as EITHER ferritin greater than 1000mcg/L OR direct bilirubin greater than 0.4 mg/dL AND platelet count less than 250,000/microL at baseline (without vaso-occlusive crisis)

E. Any one of the below complications:

-Complication: Vaso-occlusive crises;

Eligible for hydroxyurea*: At least 3 hospital admissions in the last year.

Eligible for HSCT: More than 1 hospital admission per year while on maximal tolerated dose of hydroxyurea*

-Complication: Acute chest syndrome

Eligible for hydroxyurea*: 2 prior ACS

Eligible for HSCT: any ACS while on hydroxyurea*

*hydroxyurea at maximum tolerated dose for at least 6 months

5.1.1.2 Patients with thalassemia who have grade 2 or 3 iron overload, determined by the presence of 2 or more of the following:

* portal fibrosis by liver biopsy
* inadequate chelation history (defined as failure to maintain adequate compliance with chelation with deferoxamine initiated within 18 months of the first transfusion and administered subcutaneously for 8-10 hours at least 5 days each week)
* hepatomegaly of greater than 2cm below the costochondral margin

5.1.2 Non-disease specific:

5.1.2.1 Age greater than or equal to 18 years

5.1.2.2 Haploidentical relative donor available

5.1.2.3 Ability to comprehend and willing to sign an informed consent

5.1.2.4 Negative Beta-HCG

EXCLUSION CRITERIA:

Recipient (any of the following would exclude the subject from participating)

5.2.1 6/6 HLA-matched with or without an ABO minor mismatched sibling donor

5.2.2 ECOG performance status of 3 or more

5.2.3 Evidence of uncontrolled bacterial, viral, or fungal infections (currently taking medication and progression of clinical symptoms) within one month prior to starting the conditioning regimen. Patients with fever or suspected minor infection should await resolution of symptoms before starting the conditioning regimen.

5.2.4 Major anticipated illness or organ failure incompatible with survival from PBSC transplant

5.2.5 Pregnant or lactating

5.2.6 Major ABO mismatch

INCLUSION CRITERIA:

Donor

5.3.1 Haploidentical relative donor

5.3.2 Weight greater than or equal to 20 kg (insofar that the weight difference between recipient and donor does not exceed a reasonable likelihood of being able to obtain an adequate cell dose from the donor within two aphereses)

5.3.3 Fit to receive filgrastim (G-CSF) and to give peripheral blood stem cells (blood counts and blood pressure within DTM standards)

5.3.4 No history of congestive heart failure or unstable angina, and no history of stroke)

5.3.4 Ability to comprehend and willing to sign an informed consent; assent obtained from minors

EXCLUSION CRITERIA:

Donor: (any of the following would exclude the donor from participating)

5.4.1 Pregnant or lactating

5.4.2 HIV positive

5.4.3 Hemoglobin S greater than or equal to 50 percent, or beta

thalassemia intermedia

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2009-12-14 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2026-09-10 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Courtney D Fitzhugh, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Fitzhugh CD, Hsieh MM, Taylor T, Coles W, Roskom K, Wilson D, Wright E, Jeffries N, Gamper CJ, Powell J, Luznik L, Tisdale JF. Cyclophosphamide improves engraftment in patients with SCD and severe organ damage who undergo haploidentical PBSCT. Blood Adv. 2017 Apr 19;1(11):652-661. doi: 10.1182/bloodadvances.2016002972. eCollection 2017 Apr 25. PMID 29296707
- [Derived] Leonard A, Furstenau D, Abraham A, Darbari DS, Nickel RS, Limerick E, Fitzhugh C, Hsieh M, Tisdale JF. Reduction in vaso-occlusive events following stem cell transplantation in patients with sickle cell disease. Blood Adv. 2023 Jan 24;7(2):227-234. doi: 10.1182/bloodadvances.2022008137. PMID 36240296
- [Derived] Bhat DK, Olkhanud PB, Gangaplara A, Seifuddin F, Pirooznia M, Biancotto A, Fantoni G, Pittman C, Francis B, Dagur PK, Saxena A, McCoy JP, Pfeiffer RM, Fitzhugh CD. Early Myeloid Derived Suppressor Cells (eMDSCs) Are Associated With High Donor Myeloid Chimerism Following Haploidentical HSCT for Sickle Cell Disease. Front Immunol. 2021 Nov 30;12:757279. doi: 10.3389/fimmu.2021.757279. eCollection 2021. PMID 34917079
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2009-H-0225.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 23 adults underwent non-myeloablative haplo-HSCT at the National Institutes of Health (NIH) from December 2009 through September 2015.
Groups:
- PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy): Patients received a regimen consisting of alemtuzumab, 400 cGy total body irradiation (TBI), sirolimus, and no posttransplant cyclophosphamide (PT-Cy).
- PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy): Patients received a regimen consisting of alemtuzumab, 400 cGy total body irradiation (TBI), sirolimus, and 50 mg/kg posttransplant cyclophosphamide (PT-Cy).
- PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy): Patients received a regimen consisting of alemtuzumab, 400 cGy total body irradiation (TBI), sirolimus, and 100 mg/kg posttransplant cyclophosphamide (PT-Cy).
Period: Overall Study
Arm/Group | PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy) | PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy) | PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy)
Started | 3 | 8 | 12
Completed | 3 | 7 | 12
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy) | PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy) | PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy) | Total
Number analyzed (Participants) | 3 | 8 | 12 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 8 | 12 | 23
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 5 | 9
  Male | 1 | 6 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 3 | 7 | 11 | 21
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 6 | 11 | 20
  White | 0 | 2 | 0 | 2
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Patients With Donor Type Hemoglobin
Description: Percentage of patients post transplant with sustained donor type hemoglobin on hemoglobin electrophoresis
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy) | PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy) | PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy)
Number analyzed (Participants) | 3 | 8 | 12
Participants | 0 | 3 | 6

2. Secondary Outcome: Chimeric Value That is Required to Maintain Graft Survival and Hematologic Normalcy.
Description: Define the level of chimerism required to maintain graft survival and hematologic normalcy. Hematologic normalcy may be defined as: being free from sickle cell disease.
  The chimeric status of patients will be measured on days +14 (or when subject starts to engraft), +30, +60 and +100, and periodically after day +100, by microsatellite analysis of the peripheral blood.
  Engraftment of donor cells was assessed with the use of methods that detect informative polymorphisms in regions known to contain short tandem repeats. Peripheral-blood CD3+ T cells and CD14+CD15+ myeloid cells were selected for analysis with the use of immunomagnetic beads (Dynal).
Time Frame: Up to Year 5
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy) | PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy) | PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy)
Number analyzed (Participants) | 3 | 8 | 12
Participants
  Greater than or Equal to 20% Chimerism with hematologic normalcy | 0 | 2 | 6
  Less than or Equal to 20% Chimerism with no hematologic normalcy | 3 | 6 | 6

3. Secondary Outcome: Number of Participants Who Developed Acute GVHD Grades I, II, III, IV
Description: Number of participants who developed Acute Graft vs Host Disease (GVHD) Grades I, II, III, IV as defined by CIMBTR criteria for Organ Stages of Acute GVHD.
  Grades are defined as:
  Grade I: Skin = Maculopapular rash< 25% of body surface area (BSA); Liver = Total Bilirubin 2-3 mg/dL; Lower GI = stool output/day is 500-999 mL/day.
  Grade II: Skin = rash on 25-50 percent body surface area; Liver = Total Bilirubin 3.1-6.0 mg/dL; Lower GI = Diarrhea 1001-1500 mL/day.
  Grade III: Skin = Rash on >50% of body surface; Liver = Total Bilirubin 6.1 - 15.0 mg/dL; Lower GI = Diarrhea > 1500 mL/day.
  Grade IV: Skin = Generalized erythroderma plus bullous formation; Liver = Total Bilirubin >15 mg/dL; Lower GI = Severe abdominal pain with or without ileus.
  Grade I GVHD is characterized as mild disease, grade II GVHD as moderate, grade III as severe, and grade IV life-threatening.
Time Frame: Day100
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy) | PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy) | PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy)
Number analyzed (Participants) | 3 | 8 | 12
Participants
  Grade I acute GvHD | 0 | 1 | 1
  Grade II acute GvHD | 0 | 0 | 0
  Grade III acute GvHD | 0 | 0 | 0
  Grade IV acute GvHD | 0 | 0 | 0

4. Secondary Outcome: Number of Participants Who Developed Limited Chronic GVHD
Description: Number of incidences of participants who developed Limited Chronic Graft vs Host Disease (GVHD).
  Limited disease is characterized by localized skin involvement and/or evidence of hepatic dysfunction.
  Limited disease is associated with a favorable outcome without systemic therapy, while extensive disease patients have an unfavorable outcome.
Time Frame: Year 5
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy) | PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy) | PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy)
Number analyzed (Participants) | 3 | 8 | 12
Participants | 0 | 0 | 1

5. Secondary Outcome: Number of Participants Who Develop Extensive GVHD
Description: Number of participants with extensive, Chronic Graft vs Host Disease (GVHD). Extensive chronic GVHD is defined as GVHD occurring after day 100 that did not meet the definition of limited chronic GVHD.
  Extensive disease presents either with generalized skin involvement, or with localized skin involvement or hepatic dysfunction plus at least one of the following:
  * Liver histology showing chronic progressive hepatitis, bridging necrosis, or cirrhosis
  * Involvement of the eye (Schirmer's test with less than 5 mm wetting) (see "Diagnosis and classification of Sjögren's syndrome")
  * Involvement of minor salivary glands or oral mucosa (as demonstrated on labial or mucosal biopsy specimen)
  * Involvement of any other target organ
Time Frame: Year 5
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy) | PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy) | PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy)
Number analyzed (Participants) | 3 | 8 | 12
Participants | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Disease-free Survival
Description: Number of participants with disease-free survival, as defined by: alive and free acute complications related to sickle cell disease.
Time Frame: Year 5
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy) | PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy) | PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy)
Number analyzed (Participants) | 3 | 8 | 12
Participants | 0 | 2 | 6

7. Secondary Outcome: Number of Participants Overall Survival
Description: Number of participants overall survival by year 5
Time Frame: Up to Year 5
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy) | PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy) | PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy)
Number analyzed (Participants) | 3 | 8 | 12
Participants
  Alive | 1 | 7 | 11
  Deceased | 2 | 1 | 1

8. Secondary Outcome: Number of Participants With Graft Failure
Description: Number of participants with graft failure by year 5. Graft failure is defined by return of sickle cell disease.
Time Frame: Up to Year 5
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy) | PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy) | PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy)
Number analyzed (Participants) | 3 | 8 | 12
Participants | 3 | 6 | 6

9. Secondary Outcome: Number of Participants That Experienced a Transplant-related Mortality
Description: Number of participants that experienced a transplant related mortality, as defined as death from causes other than relapse (GVHD, toxicity, infection, other and unknown causes).
Time Frame: Year 1
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy) | PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy) | PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy)
Number analyzed (Participants) | 3 | 8 | 12
Participants | 0 | 1 | 0

10. Secondary Outcome: Number of Stem Cell Transplant Participants That Experienced Rejection at Each Dose of Post-transplant Cyclophosphamide
Description: Number of stem cell transplant participants that experienced rejection at each dose of post-transplant cyclophosphamide. Determine whether post-transplant cyclophosphamide is required and will reduce the incidence and severity of regimen failure.
Time Frame: Year 5
Measure: Count of Participants; unit: Participants
Arm/Group | PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy) | PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy) | PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy)
Number analyzed (Participants) | 3 | 8 | 12
Participants
  No post-transplant cyclophosphamide | 3 | 0 | 0
  50 mg/kg posttransplant cyclophosphamide | 0 | 6 | 0
  100 mg/kg posttransplant cyclophosphamide | 0 | 0 | 6

11. Secondary Outcome: Participants Who Engrafted or Rejected and Type of Haploidentical Donors
Description: Determine whether specific haploidentical donors (i.e. parent versus sibling versus child) will decrease the incidence of regimen failure
Time Frame: Up to Year 5
Population: Participants with Sickle Cell Disease who survived beyond 6 months (participants with beta-thalassemia were excluded).
Measure: Count of Participants; unit: Participants
Groups:
- Participants Who Engrafted Following Stem Cell Transplant; Participants Who Rejected Engraftment Following Stem Cell Transplant: Engrafted participants received a regimen consisting of alemtuzumab, 400 cGy total body irradiation (TBI), sirolimus, and posttransplant cyclophosphamide (PT-Cy) from 0 to 100 mg/kg, followed by infusion of haploidentical stem cells.
Arm/Group | Participants Who Engrafted Following Stem Cell Transplant | Participants Who Rejected Engraftment Following Stem Cell Transplant
Number analyzed (Participants) | 8 | 12
Participants
  Father | 0 | 1
  Mother | 3 | 6
  Brother | 2 | 1
  Sister | 3 | 3
  Son | 0 | 1

ADVERSE EVENTS:
Time Frame: 5 year
Description: Adverse events will be solicited from participant through questions from study personnel and information volunteered by the participant.
Arm/Group | PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy) | PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy) | PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy)
All-Cause Mortality (participants affected / at risk) | 2/3 | 1/8 | 1/12
Serious Adverse Events (participants affected / at risk) | 3/3 | 7/8 | 11/12
Other Adverse Events (participants affected / at risk) | 0/3 | 0/8 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PBSC Transplant With no Post-transplant Cyclophosphamide (PT-Cy) (N=3) | PBSC Transplant With 50 mg/kg Post-transplant Cyclophosphamide (PT- Cy) (N=8) | PBSC Transplant With 100 mg/kg Post-transplant Cyclophosphamide (PT- Cy) (N=12)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Myelodysplastic syndrome (Blood and lymphatic system disorders) | 1 | 0 | 1
Sickle cell anemia with crisis (Blood and lymphatic system disorders) | 0 | 0 | 2
Cardiovascular disorder (Cardiac disorders) | 0 | 1 | 1
Syncope (Cardiac disorders) | 0 | 0 | 2
Ventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1
Upper gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Device related infection (General disorders) | 0 | 0 | 1
Device related thrombosis (General disorders) | 1 | 1 | 0
Extravasation (General disorders) | 0 | 1 | 0
Inflammation (General disorders) | 0 | 1 | 1
Pain (General disorders) | 1 | 2 | 4
Hepatic hemorrhage (Hepatobiliary disorders) | 0 | 0 | 1
Portal hypertension (Hepatobiliary disorders) | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 4 | 6
Infective Myositis (Infections and infestations) | 0 | 0 | 1
Lung infection (Infections and infestations) | 1 | 0 | 2
Sepsis (Infections and infestations) | 0 | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 2
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 1
Seizure (Nervous system disorders) | 0 | 0 | 1
Ectopic pregnancy while on Mycophenolate Mofetil (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pulmonary Hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Embolism (Vascular disorders) | 0 | 1 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Bacteremia (Infections and infestations) | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 0 | 1
Esophageal varices (Gastrointestinal disorders) | 0 | 0 | 1
Liposarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1
Electrolyte imbalance (General disorders) | 0 | 0 | 1
Intracranial hemmorhage (Nervous system disorders) | 0 | 0 | 1
Benign Neuroendocrine Tumor (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Noncardiac Chest Pain (General disorders) | 0 | 0 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Norovirus (Infections and infestations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/91/NCT00977691/Prot_SAP_000.pdf